CLINICAL TRIAL: NCT03238898
Title: Botulinum Toxin for Muscle Cramps in Diabetic Patients With Diabetic Neuropathy
Brief Title: Botulinum Toxin for Cramps in Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Presidio Ospedaliero Garibaldi-Centro (Other)
Responsible Party: Principal Investigator, Domenico Antonio Restivo, Dr, Presidio Ospedaliero Garibaldi-Centro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: btx for cramps
Record Dates: First submitted 2017-06-09; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Muscle Cramps Aggravated; Diabetes Mellitus
Keywords: muscle cramps; diabetic neuropathy; botulinum toxin
MeSH Terms: conditions — Diabetes Mellitus; Muscle Cramp; Diabetic Neuropathies | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, double-blind and placebo-controlled study
Who Masked: Participant
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- botulinum toxin type A (Active Comparator): Botulinum toxin type A (100 or 30 units) was injected for each side into the gastrocnemious or the small flexor foot muscles, respectively, according to the predominance of leg or foot cramps.
  Interventions: Drug: Botulinum toxin type A
- Normal saline (Placebo Comparator): The same dosage as the active group, but with normal saline alone were injected into the gastrocnemious or the small flexor foot muscles, respectively, according to the predominance of leg or foot cramps.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Botulinum toxin type A — botulinum toxin type A injections
  Botulinum toxin type A (100 or 30 units) was injected for each side into the gastrocnemious or the small flexor foot muscles, respectively, according to the predominance of leg or foot cramps.
  Arms: botulinum toxin type A
Other: Normal saline — Normal saline injections
  The same dosage as the active group, but with normal saline alone were injected into the gastrocnemious or the small flexor foot muscles, respectively, according to the predominance of leg or foot cramps.
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
Objective: previous studies suggest that botulinum toxin A (BoNT/A) can reduce muscle hyperactivity.

Research Design and Methods: a single-center, double-blind and placebo-controlled study investigating the efficacy and safety of BoNT/A intramuscular injection for treating calf or foot cramps refractory to common pharmacological drugs in patients with diabetic peripheral neuropathy. Fifty patients were subdivided in two matched groups (cases and controls) and BoNT/A (100 or 30 units) was injected for each side into the gastrocnemious or the small flexor foot muscles, respectively, according to the predominance of leg or foot cramps. Responders were evaluated again with a second BoNT/A administration.

The changes of pain intensity (primary outcome) and the changes in cramp frequency, the and the Cramp Severity Scale (CSS) were evaluated over the course of 20 weeks after BoNT/A administration.

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, placebo-controlled prospective study.

A consecutive series of 303 out-patients with type 2 diabetes was screened for muscle cramps.Patients were asked to report in a questionnaire the frequency, localization, intensity and time of the day of cramps. Out of these 303 diabetic patients with cramps, fifty patients satisfied the inclusion/exclusion criteria and entered the study.

Cramp Evaluation

a) Clinical evaluation All patients completed a baseline diary in the week before treatment. Every day the number of muscle cramp episodes was reported three times a day and the intensity of pain was rated on a scale 0 to 10, with 0 indicating no pain and 10 indicating "the worst pain imaginable" (Brief Pain Inventory-Modified Short Form, BPI-MSF, point 1). Daily data in this pre-treatment week were averaged and considered "basal" values. A similar daily diary, reporting the number of pain episodes, their intensity, time of the day and duration (less or more than 1 min) was kept throughout the study for the three days before each control visit.

The severity of cramps interference on daily life was graded according to the functional scale Cramp Severity Score (CSS): 0= no cramps; 1= occasional day or night cramps not interfering with daily activities or with nocturnal sleep; 2= frequent muscle cramps triggered by muscle exercise not significantly interfering with daily activity or with nocturnal sleep; 3= continuous or subcontinuous muscle cramps limiting daily activities or nocturnal sleep; 4= continuous cramps severely interfering with daily activities and nocturnal sleep (4).

Randomisation: patients were randomly assigned to either the treatment or control groups according to a computer-generated list. Randomization was stratified in order to match age, gender, duration of diabetes and the frequency and severity of cramp episodes in the two groups.

At time 0 each patient received four i.m. injections, two injections for each side, containing either BoNT/A (100 units diluted in 1 ml saline) or saline. The total dose, for each side, was 100 units for the gastrocnemius muscle or 30 units for the small flexor foot muscles. The calf or the foot muscles were chosen according to the patient predominant leg or foot cramps. Patients in the control group received the same volumes of normal saline in the same muscles. The injections were prepared by a research nurse and both the treating physician and the patients were left blind.

Ten visits were scheduled after initial evaluation: at weeks 1 and 2 after BoNT/A injection and, thereafter, every other week until week 16 and then at week 20. Ratings of the three days before each control visit were averaged to obtain values for each post-injection evaluation. The number of cramp episodes and cramp severity score (both self-reported in the daily diary) were obtained at 1, 4, 8, 12, 16 and 20 weeks after BoNT/A or placebo administration.

Positive response to treatment: a 30% or greater reduction of the primary outcome score.

ELIGIBILITY:
Inclusion Criteria:

* accepting to participate to the study;
* age ≥ 45 and ≤ 75 years ;
* diabetes duration > 5 years and diabetic distal symmetric neuropathy present;
* stable glycemic control with last HbA1c value <9.0% (or 75 mmol/mol);
* cramps present at rest in either calf or foot muscles or both for at least 6 months;
* occurrence of cramps at least 3 times a week in the previous three months;
* previous unsuccessful or poorly tolerated pharmacological treatment with at least two of the following drugs: carbamazepine, quinine, phenytoin, magnesium supplements, and benzodiazepines.

Exclusion Criteria:

* the presence of other neurological diseases and of nephropathy, macro-angiopathy, cirrhosis, and lumbar disc diseases or the inability to give informed consent because of cognitive impairment.
* Patients previously treated with BoNT/A for any reason were also excluded

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-27 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
pain intensity on a 0-10 severity scale | 20 weeks
  the intensity of pain was rated on a scale 0 to 10, with 0 indicating no pain and 10 indicating "the worst pain imaginable"

SECONDARY OUTCOMES:
cramp frequency | 20 weeks
  the changes in cramp frequency, the Cramp Severity Scale (CSS) were evaluated over the course of 20 weeks after BoNT/A administration
the Cramp Severity Scale (CSS) | 20 weeks
  the changes in the Cramp Severity Scale (CSS) were evaluated over the course of 20 weeks after BoNT/A administration
the Cramp Threshold Frequency (CTF) | 20 weeks
  the changes in the Cramp Threshold Frequency were evaluated over the course of 20 weeks after BoNT/A administration

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertolasi L, Priori A, Tomelleri G, Bongiovanni LG, Fincati E, Simonati A, De Grandis D, Rizzuto N. Botulinum toxin treatment of muscle cramps: a clinical and neurophysiological study. Ann Neurol. 1997 Feb;41(2):181-6. doi: 10.1002/ana.410410209. PMID 9029067